CLINICAL TRIAL: NCT03748017
Title: The Probiotic for Oral Health (PRO Health) Study
Acronym: PRO Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Renew Life Formulas Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1188050
Record Dates: First submitted 2018-10-22; First posted 2018-11-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Oral Microbiome

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled and randomized, receiving either a streptococcus-containing probiotic supplement or a placebo-control supplement.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and data evaluators will be blinded to the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Control Supplement (Placebo Comparator): 12 participants will receive a placebo-control supplement per daily oral feeding.
  Interventions: Dietary Supplement: Placebo-Control Supplement
- Streptococcus-Containing Probiotic Supplement (Active Comparator): 12 participants will receive a powdered probiotic containing 7.77 billion colony-forming units (CFU) of L. acidophilus, 8.25 billion CFU of B. lactis, and 2 billion CFU of S. salivarius bacteriocin-like inhibitory substance (BLIS) K12 per daily oral feeding.
  Interventions: Dietary Supplement: Streptococcus-Containing Probiotic Supplement

INTERVENTIONS:
Dietary Supplement: Placebo-Control Supplement — A once-daily oral dose of the placebo-control supplement will be consumed by adults for 14 consecutive days.
  Arms: Placebo-Control Supplement
Dietary Supplement: Streptococcus-Containing Probiotic Supplement — A once-daily oral dose of the streptococcus-containing probiotic supplement will be consumed by adults for 14 consecutive days.
  Arms: Streptococcus-Containing Probiotic Supplement

SUMMARY:
The PRO Health Study is a single-center, prospective, double-blind, randomized, placebo-controlled trial of streptococcus-containing supplementation in healthy adults.

DETAILED DESCRIPTION:
Upon enrollment, healthy adults will enter a 1-week lead-in period which serves as an opportunity to collect baseline saliva samples and complete daily logs. Subjects that meet eligibility criteria on Day 7 will be randomized into 1 of 2 groups, receiving either a placebo-control or a streptococcus-containing probiotic supplement. Supplementation will begin on Day 8 and will continue for a total of 14 consecutive days. Participants will be observed for an additional 2 weeks following cessation of supplementation. The total duration of the study will be approximately 5 weeks. Saliva samples will be collected on 7 occasions and participants will be asked to complete questionnaires and daily diet and health logs throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 21-45 years of age;
* BMI between 18-30;
* No history of infectious disease; heart, metabolic, autoimmune endocrine, liver, or kidney diseases; GI related conditions such as malabsorption disease, Crohn's disease, colitis, inflammatory bowel disease; Type 1 or 2 diabetes mellitus, any type of cancer, heart disease;
* Practices good oral hygiene according to the American Dental Association with brushing teeth between 1-2 times per day;
* Willingness to only use the study toothpaste to brush or clean teeth and refrain from using any other oral-care products such as other toothpaste, mouthwash, rinses and breath-sprays during the five-week study period;
* Willingness to limit consumption of raw onions or garlic and fermented foods such as sauerkraut, pickles, miso, and kimchi during the five-week study period;
* Non-alcohol consumers or those who consume alcohol in moderation defined as having up to 1 drink per day for women and up to 2 drinks per day for men;
* Willingness to avoid binge drinking during the study period defined by the Centers for Disease Control and Prevention as: This pattern of drinking usually corresponds to 5 or more drinks on a single occasion for men or 4 or more drinks on a single occasion for women, generally within about 2 hours;
* Willingness to refrain from drinking any alcohol within 24 hours of each saliva sample collection;
* Willingness to refrain from using illicit drugs during the five-week study;
* Willingness to refrain from using tobacco (smoking or chewing) or smoking marijuana during the five-week study period;
* Willingness to refrain from intake of probiotics, kombucha, or yogurt during the five-week study period;
* Willingness to refrain from consuming more than 1 package of sugary candy and from chewing more than 1 package of chewing gum during the five-week study period;
* Willingness to refrain from having any non-emergency, elective oral surgeries, dental procedures or dental teeth cleanings during the five-week study period.

Exclusion Criteria:

* Currently pregnant or plans to become pregnant several weeks prior to enrollment and during the five-week study period;
* History of periodontal disease, or gingivitis;
* Dental trauma or injury to the teeth and/or periodontium (gums, periodontal ligament, alveolar bone), and nearby soft tissues such as the lips, tongue within the past 4 weeks;
* Any oral surgery or intensive procedures made to the oral cavity (such as fillings, wisdom tooth extraction, root canal, dental implants, etc.) within the past 4 weeks;
* Routine dental cleaning within the past 4 weeks;
* Use of probiotics, kombucha, or yogurt/kefir within the past 7 days of enrollment;
* Use of probiotics containing S. salivarius within the past 8 weeks of enrollment;
* Use of oral or IV antibiotics within the past 8 weeks of enrollment;
* Consumption of more than one package of sugary candy (hard candy, gummy candy, mints, etc.) per day;
* Use of more than one package of chewing gum (sugary or sugarless) per day;
* Use of mouthwashes, mouth-rinses or breath-sprays more than three times per day;
* Current tobacco (smoking or chewing) or E-cigarette users or individuals who quit using less than one year before enrolling in the study;
* Frequent marijuana smoking or vaping, or use of other illicit drugs (must be no more than 12 times within the past year and no more than once per month);
* Marijuana smoking or vaping or use of other illicit drugs within the past 4 weeks;
* Excessive alcohol drinkers: For men, heavy drinking is typically defined as consuming 15 drinks or more per week. For women, heavy drinking is typically defined as consuming 8 drinks or more per week;
* Individuals who live within the same household or who are in intimate relationships with current or past study participants (to avoid horizontal transfer of the oral microbiome);
* Anyone the investigator feels isn't an applicable participant.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Oral Streptococci levels in adults at 22 days - difference between S. Salivarius and placebo | 22 Days
  The difference in levels of oral Streptococci between a streptococcus-containing probiotic supplement (e.g., S. salivarius K12) and placebo-control supplement on Day 22.

SECONDARY OUTCOMES:
Oral Streptococcus levels | Change from baseline, days 10, 14, 22, 28, 36
  The difference in levels of Streptococci upon intake of a streptococcus-containing probiotic supplement (e.g., S. salivarius K12) before, during and after the intervention compared with a placebo-control supplement.
Oral microbiome | Change from baseline, days 10, 14, 22, 28, 36
  The difference in the salivary microbiome before, during and after intake of a streptococcus-containing probiotic supplement (e.g., S. salivarius K12) and placebo-control supplement.
Number of stools per day | Change from baseline, days 10, 14, 22, 28, 36
  The relationship between supplementation and number of stools per day.
Changes in stool consistency | Change from baseline, days 10, 14, 22, 28, 36
  The relationship between supplementation and number of stools per day, rated using the Bristol Stool Scale.
Changes in stool firmness | Change from baseline, days 10, 14, 22, 28, 36
  The relationship between supplementation and number of stools per day, rated using a continuous scale of 1 to 10 (1 = extremely watery, almost entirely liquid to 10 = extremely hard, difficult to pass).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horz HP, Meinelt A, Houben B, Conrads G. Distribution and persistence of probiotic Streptococcus salivarius K12 in the human oral cavity as determined by real-time quantitative polymerase chain reaction. Oral Microbiol Immunol. 2007 Apr;22(2):126-30. doi: 10.1111/j.1399-302X.2007.00334.x. PMID 17311636
- [Background] Upton M, Tagg JR, Wescombe P, Jenkinson HF. Intra- and interspecies signaling between Streptococcus salivarius and Streptococcus pyogenes mediated by SalA and SalA1 lantibiotic peptides. J Bacteriol. 2001 Jul;183(13):3931-8. doi: 10.1128/JB.183.13.3931-3938.2001. PMID 11395456
- [Background] Ross KF, Ronson CW, Tagg JR. Isolation and characterization of the lantibiotic salivaricin A and its structural gene salA from Streptococcus salivarius 20P3. Appl Environ Microbiol. 1993 Jul;59(7):2014-21. doi: 10.1128/aem.59.7.2014-2021.1993. PMID 8357242
- [Background] Cosseau C, Devine DA, Dullaghan E, Gardy JL, Chikatamarla A, Gellatly S, Yu LL, Pistolic J, Falsafi R, Tagg J, Hancock RE. The commensal Streptococcus salivarius K12 downregulates the innate immune responses of human epithelial cells and promotes host-microbe homeostasis. Infect Immun. 2008 Sep;76(9):4163-75. doi: 10.1128/IAI.00188-08. Epub 2008 Jul 14. PMID 18625732
- [Background] Di Pierro F, Adami T, Rapacioli G, Giardini N, Streitberger C. Clinical evaluation of the oral probiotic Streptococcus salivarius K12 in the prevention of recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes in adults. Expert Opin Biol Ther. 2013 Mar;13(3):339-43. doi: 10.1517/14712598.2013.758711. Epub 2013 Jan 4. PMID 23286823
- [Background] Di Pierro F, Colombo M, Zanvit A, Rottoli AS. Positive clinical outcomes derived from using Streptococcus salivarius K12 to prevent streptococcal pharyngotonsillitis in children: a pilot investigation. Drug Healthc Patient Saf. 2016 Nov 21;8:77-81. doi: 10.2147/DHPS.S117214. eCollection 2016. PMID 27920580
- [Background] Di Pierro F, Donato G, Fomia F, Adami T, Careddu D, Cassandro C, Albera R. Preliminary pediatric clinical evaluation of the oral probiotic Streptococcus salivarius K12 in preventing recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes and recurrent acute otitis media. Int J Gen Med. 2012;5:991-7. doi: 10.2147/IJGM.S38859. Epub 2012 Nov 30. PMID 23233809
- [Background] Di Pierro F, Colombo M, Giuliani MG, Danza ML, Basile I, Bollani T, Conti AM, Zanvit A, Rottoli AS. Effect of administration of Streptococcus salivarius K12 on the occurrence of streptococcal pharyngo-tonsillitis, scarlet fever and acute otitis media in 3 years old children. Eur Rev Med Pharmacol Sci. 2016 Nov;20(21):4601-4606. PMID 27874935
- [Background] Burton JP, Chilcott CN, Tagg JR. The rationale and potential for the reduction of oral malodour using Streptococcus salivarius probiotics. Oral Dis. 2005;11 Suppl 1:29-31. doi: 10.1111/j.1601-0825.2005.01084.x. PMID 15752094
- [Background] Burton JP, Chilcott CN, Moore CJ, Speiser G, Tagg JR. A preliminary study of the effect of probiotic Streptococcus salivarius K12 on oral malodour parameters. J Appl Microbiol. 2006 Apr;100(4):754-64. doi: 10.1111/j.1365-2672.2006.02837.x. PMID 16553730
- [Background] Bourdichon F, Casaregola S, Farrokh C, Frisvad JC, Gerds ML, Hammes WP, Harnett J, Huys G, Laulund S, Ouwehand A, Powell IB, Prajapati JB, Seto Y, Ter Schure E, Van Boven A, Vankerckhoven V, Zgoda A, Tuijtelaars S, Hansen EB. Food fermentations: microorganisms with technological beneficial use. Int J Food Microbiol. 2012 Mar 15;154(3):87-97. doi: 10.1016/j.ijfoodmicro.2011.12.030. Epub 2011 Dec 31. PMID 22257932
- [Background] Authority, E.F.S., Introduction of a Qualified Presumption of Safety (QPS) approach for assessment of selected microorganisms referred to EFSA-Opinion of the Scientific Committee. EFSA Journal, 2007. 5(12): p. 587.
- [Background] Mogensen, G., et al., Inventory of microoganisms with a documented history of use in food. 2002.